CLINICAL TRIAL: NCT06659120
Title: Fremanezumab for the Prevention of Menstrually-related Migraine Attacks - a Prospective, Observational Study According to Routine Neurological Care in Switzerland
Brief Title: Fremanezumab for the Prevention of Menstrually-related Migraine Attacks
Acronym: FROMM
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00388
Record Dates: First submitted 2024-08-12; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Menstrual Migraine
MeSH Terms: interventions — fremanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with menstrually-related migraine attacks: * Premenopausal women of 18 years of age or older.
  * Women with a regular cycle 21-32 days.
  * The patient has a diagnosis of chronic or episodic migraine.
  * Women suffering from migraine with or without aura according to International Headache Society (IHS) Classification (ICHD-3 code A1.1.2 or A1.2.0.2) for at least one year.
  * Women suffering of at least 2 days of menstrually-related migraine per period on average in the last three periods (baseline measurements and inclusion criteria).
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Initiation of anti-CGRP mAb (fremanezumab) treatment according to the Summary of Product Characteristics (SmPC) during clinical routine as a treatment of their physician (no study-specific intervention). This means that patients have to fulfil criteria for treatment with anti-CGRP mAbs in Switzerland, i.e. they have at least 8 days of migraine per month in the last three months.

SUMMARY:
The goal of this observational study is to compare, in real-world clinical practice, the effect of fremanezumab on menstrual migraine to the effect of fremanezumab on non-perimenstrual attacks. The main question it aims to answer is, if menstrually-related migraine attacks respond equally well to anti-CGRP mAb treatment with fremanezumab as non-menstrually-related attacks.

Participants diagnosed with episodic or chronic migraine with menstrually-related migraine with or without aura and treated with fremanzumab according to the SmPC will be required to maintain a headache diary over at least 3 months prior to and 6 months after fremanezumab initiation.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women of 18 years of age or older.
* Women with a regular cycle 21-32 days.
* The patient has a diagnosis of chronic or episodic migraine.
* Women suffering from migraine with or without aura according to International Headache Society (IHS) Classification (ICHD-3 code A1.1.2 or A1.2.0.2) for at least one year.
* Women suffering of at least 2 days of menstrually-related migraine per period on average in the last three periods (baseline measurements and inclusion criteria).
* The patient has been maintaining a daily headache diary as part of her routine disease management per her treating physician and has 3 months headache diary data prior to baseline/ treatment initiation. Notes: The patient's headache diary captures information on each headache day, headache duration, headache severity, medication intake, each day of menstrual bleeding, pain intensity of symptoms associated with the menstrual bleeding and symptoms of endometriosis (if present): dysmenorrhoea, dyschezia, dyspareunia, dysuria.
* The patient understands and is willing to keep records in their headache diary for the course of the study.
* Initiation of anti-CGRP mAb (fremanezumab) treatment according to the Summary of Product Characteristics (SmPC) during clinical routine as a treatment of their physician (no study-specific intervention). This means that patients have to fulfil criteria for treatment with anti-CGRP mAbs in Switzerland, i.e. they have at least 8 days of migraine per month in the last three months.
* The patient has signed the informed consent.

Exclusion Criteria:

* Patients with pure menstrual migraine.
* The patient is treated with another anti-CGRP mAb.
* The patient is not treated with fremanezumab according to the SmPC.
* The patient is being treated with another anti-CGRP-based preventive migraine medication within 6 months of enrolment.
* The patient is participating in an interventional clinical trial in EM or CM.
* Change of hormone therapy during study treatment.
* Progestin-only contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premenopausal women ≥18 years of age, diagnosed with episodic or chronic migraine, with menstrually-related migraine with or without aura according to IHS Classification (ICHD-3 code A1.1.2 or A1.2.0.2)*, and have been prescribed fremanezumab according to the SmPC as a treatment decision of their physician and enrollment in this study at baseline.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of migraine days per month | 6 months
  Difference in relative reduction of migraine days per month between menstrually-related and non-menstrual migraine days at follow-up (months 4 to 6 after initiation of anti-CGRP mAb) compared to baseline (months -3 to -1 prior to initiation).

SECONDARY OUTCOMES:
Change of disability score MIDAS in points | 6 months
  Change from baseline in disability score, as measured by the Migraine Disability Assessment (MIDAS) questionnaire, at month 6.
Change of headache-related disability score HIT-6 in points | 6 months
  Headache-related disability score, as measured by the HIT-6, at month 6.
Migraine-specific quality of life in MSQ score in points | 6 months
  Migraine-specific quality of life, as measured by the MSQ version 2.1, at month 6.
Anxiety in GAD-7 score, in points | 6 months
  Change from baseline in anxiety (GAD-7).
Depression in PHQ-8 score, in points | 6 months
  Change from baseline in depression (PHQ-8).
Change of fatigue assessed by FSS in points | 6 months
  Change from baseline in sleep questionnaires at month 6 (Fatigue Severity Scale (FSS), Epworth Sleepiness Scale (ESS) and Insomnia Severity Index (ISI)).
Endometriosis symptoms | 6 months
  Change from baseline in number of days per month and intensity with typical symptoms of endometriosis (dysmenorrhoea, dyschezia, dysuria and dyspareunia) in women who have menstrually-related migraine and endometriosis (subgroup) at follow-up (months 4 to 6 after initiation of anti-CGRP mAb) compared to baseline (months -3 to -1 prior to initiation). (Headache diary).
Hormonal treatment | 6 months
  Change from baseline in number of migraine days in patients with and without concomitant hormonal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph J Schankin, Prof, Principal Investigator — Inselspital, Department of Neurology, Bern
Locations (1):
- Department of Neurology, Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Russell MB, Rasmussen BK, Thorvaldsen P, Olesen J. Prevalence and sex-ratio of the subtypes of migraine. Int J Epidemiol. 1995 Jun;24(3):612-8. doi: 10.1093/ije/24.3.612. PMID 7672904
- [Background] Celentano DD, Linet MS, Stewart WF. Gender differences in the experience of headache. Soc Sci Med. 1990;30(12):1289-95. doi: 10.1016/0277-9536(90)90309-g. PMID 2367875
- [Background] MacGregor EA, Hackshaw A. Prevalence of migraine on each day of the natural menstrual cycle. Neurology. 2004 Jul 27;63(2):351-3. doi: 10.1212/01.wnl.0000133134.68143.2e. PMID 15277635
- [Background] Chalmer MA, Kogelman LJA, Ullum H, Sorensen E, Didriksen M, Mikkelsen S, Dinh KM, Brodersen T, Nielsen KR, Bruun MT, Banasik K, Brunak S, Erikstrup C, Pedersen OB, Ostrowski SR, Olesen J, Hansen TF. Population-Based Characterization of Menstrual Migraine and Proposed Diagnostic Criteria. JAMA Netw Open. 2023 May 1;6(5):e2313235. doi: 10.1001/jamanetworkopen.2023.13235. PMID 37184838
- [Background] Calhoun A, Ford S. Elimination of menstrual-related migraine beneficially impacts chronification and medication overuse. Headache. 2008 Sep;48(8):1186-93. doi: 10.1111/j.1526-4610.2008.01176.x. PMID 18819179
- [Background] Sevivas H, Fresco P. Treatment of resistant chronic migraine with anti-CGRP monoclonal antibodies: a systematic review. Eur J Med Res. 2022 Jun 4;27(1):86. doi: 10.1186/s40001-022-00716-w. PMID 35659086
- [Background] Ornello R, Frattale I, Caponnetto V, De Matteis E, Pistoia F, Sacco S. Menstrual Headache in Women with Chronic Migraine Treated with Erenumab: An Observational Case Series. Brain Sci. 2021 Mar 13;11(3):370. doi: 10.3390/brainsci11030370. PMID 33805838
- [Background] Verhagen IE, de Vries Lentsch S, van der Arend BWH, le Cessie S, MaassenVanDenBrink A, Terwindt GM. Both perimenstrual and nonperimenstrual migraine days respond to anti-calcitonin gene-related peptide (receptor) antibodies. Eur J Neurol. 2023 Jul;30(7):2117-2121. doi: 10.1111/ene.15794. Epub 2023 Apr 6. PMID 36941533
- [Background] van Casteren DS, Verhagen IE, van der Arend BWH, van Zwet EW, MaassenVanDenBrink A, Terwindt GM. Comparing Perimenstrual and Nonperimenstrual Migraine Attacks Using an e-Diary. Neurology. 2021 Oct 26;97(17):e1661-e1671. doi: 10.1212/WNL.0000000000012723. Epub 2021 Sep 7. PMID 34493613
- [Background] Pavlovic JM, Paemeleire K, Gobel H, Bonner J, Rapoport A, Kagan R, Zhang F, Picard H, Mikol DD. Efficacy and safety of erenumab in women with a history of menstrual migraine. J Headache Pain. 2020 Aug 3;21(1):95. doi: 10.1186/s10194-020-01167-6. PMID 32746775
- [Background] Silvestro M, Orologio I, Bonavita S, Scotto di Clemente F, Fasano C, Tessitore A, Tedeschi G, Russo A. Effectiveness and Safety of CGRP-mAbs in Menstrual-Related Migraine: A Real-World Experience. Pain Ther. 2021 Dec;10(2):1203-1214. doi: 10.1007/s40122-021-00273-w. Epub 2021 Jun 9. PMID 34106431